CLINICAL TRIAL: NCT04533243
Title: Opioid Titration With 12.5 ug/h Fentanyl Transdermal Patch vs Orally Morphine for Opioid-naïve Patients With Moderate Cancer Pain: A Prospective, Randomized, Controlled, Multi-center, Phase III Trial
Brief Title: Opioid Titration With 12.5 ug/h Fentanyl Transdermal Patch vs Orally Morphine for Opioid-naïve Patients With Moderate Cancer Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYLT-19
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Opioid, Moderate Cancer Pain, Transdermal Fentanyl, 12.5ug/h, Opioid-naive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2.5ug/h transdermal fentanyl (Experimental)
  Interventions: Drug: 2.5ug/h transdermal fentanyl
- Oral immediate-released morphine (Active Comparator)
  Interventions: Drug: Oral immediate-released morphine

INTERVENTIONS:
Drug: 2.5ug/h transdermal fentanyl — 2.5ug/h transdermal fentanyl administers for opioid-naive patients with moderate cancer pain very 3 days
  Arms: 2.5ug/h transdermal fentanyl
Drug: Oral immediate-released morphine — 5mg immediate-released morphine every 4 hours, double dose before sleep.
  Arms: Oral immediate-released morphine

SUMMARY:
Opioid is recommended for moderate cancer pain in WHO 3-step analgesic ladder. Transdermal administration of the strong opioid fentanyl was originally developed for patients unable to swallow analgesics because of malignancies in the head and neck region or the gastrointestinal tract, painful lesions in the mouth, or periods of nausea, vomiting, or bowel obstruction. The EMA recognizes that in exceptional clinical circumstances, the 12 μg/h fentanyl patch could be considered. To our knowledge, there is not a phase III trial to explore the efficacy and safety of 12 μg/h fentanyl patch in opioid-naive patients with moderate cancer pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old or more;
2. ECOG PS ≤3 ;
3. Opioid tolerance not moderate pain patients (4≤ NRS ≤6 on 11 points, 0 no pain, 10 most pain);
4. No taking strong opioids for the last 30 days;
5. Estimated life expectancy of at least 3 months;
6. Ability to communicate effectively with the study personnel about the nature of their pain;
7. Ability to complete a diary;
8. Cancer pain is expected to be relatively stable and last for more than 48 hours;
9. The patient understands the research process, agrees to participate in the trial, cooperates with the treatment and visit plan, and signs an informed consent form.

Exclusion Criteria:

1. Known allergy to any ingredient in both fentanyl and morphine;
2. No cancer associated pain or the pain of unknown cause, such as osteoarthritis pain, acute abdominal pain;
3. Primary tumors or metastases in the brain;
4. An active skin disease that precluded application of the transdermal system;
5. Anti-cancer therapy (radiotherapy, chemotherapy, targeted therapy, etc.) is used during the study period, and the treatment has an impact on the analgesic effect or adverse reactions of analgesic drugs;
6. No bowel movement within 3 days before the screening period;
7. The patient has contraindications to the use of opioids: such as respiratory depression; head damage; paralytic intestinal obstruction; acute abdomen; chronic obstructive airway disease; pulmonary heart disease; chronic bronchial asthma; hypercapnia;
8. Used monoamine oxidase inhibitor within 1 week before randomization;
9. Any abnormal laboratory test results with obvious clinical significance, such as creatinine value ≥ 2 times the high limit of the normal value or ALT or AST ≥ 2.5 times the high limit of the normal value (for patients with liver metastases can be relaxed to ≥ 5 times the high limit of the normal value) ;
10. Patients with a history of drug abuse;
11. Patients with mental illness or cognitive impairment;
12. Pregnant or lactating women; subjects who have a pregnancy plan within 1 month after the test (including male subjects);
13. Participate in the drug trial (including the trial drug) within 3 months before the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
the number of responder patients | 12 months
  the number of responder patients is defined as patientswith a 20% reduction in pain intensity on the numerical rating scale.

IPD SHARING:
Plan to Share IPD: Undecided